CLINICAL TRIAL: NCT07321886
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy and Safety of Once Weekly Eloralintide in Adult Participants With Obesity or Overweight, Without Type 2 Diabetes
Brief Title: A Study of Eloralintide (LY3841136) in Participants With Obesity, or Overweight Without Type 2 Diabetes
Acronym: ENLIGHTEN-1
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27742; J3R-MC-YDAG (Other: Eli Lilly and Company); 2025-523657-34-00 (Other: EU CTIS)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Eloralintide Dose 1 (Experimental): Participants will receive eloralintide subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Eloralintide Dose 2 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 3 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Eloralintide Dose 4 (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Placebo (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide Dose 1; Eloralintide Dose 2; Eloralintide Dose 3; Eloralintide Dose 4
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of eloralintide in adults with obesity or overweight who do not have type 2 diabetes. The study has two phases: a main phase and an extension phase.

Participation in the main phase of the study will last about 75 weeks. Participants with prediabetes will continue in the extension phase for another 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have Body Mass Index (BMI) at screening of the following:

  * 30 kilogram per square meter (kg/m2) OR
  * 27 kg/m2 with at least one of the following weight-related health conditions at screening:

    * high blood pressure
    * dyslipidemia
    * obstructive sleep apnea, or
    * heart disease
* Have a stable body weight (<5% body weight change) for 90 days prior to screening.
* Have a history of at least one self-reported unsuccessful dietary effort to reduce body weight

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity (liposuction, cryolipolysis, or abdominoplasty allowed if performed >1 year before screening)
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity (prior device-based therapy acceptable if device removal was more than 6 months prior to screening)
* Have type 1 diabetes or type 2 diabetes
* Have had within 90 days prior to screening:

  * heart attack
  * stroke
  * coronary artery revascularization
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history or diagnosis of New York Heart Association Functional Classification Class IV congestive heart failure
* Have taken medications or alternative remedies intended for weight loss within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1980 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 64

SECONDARY OUTCOMES:
Percent Change from Baseline in Total Body Fat Mass | Baseline, Week 64
Change from Baseline in Waist Circumference | Baseline, Week 64
Percent Change from Baseline in Triglycerides | Baseline, Week 64
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 64
Time to Onset of Type 2 Diabetes (T2D) | Baseline to Week 168 and Week 191
  Time to Onset of Type 2 Diabetes (T2D) in Participants with Prediabetes at Randomization
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 64
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, Week 64
Percent Change from Baseline in Fasting Insulin | Baseline, Week 64
Percent Change from Baseline in High-Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 64
Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 64
Change from Baseline in Short Form-36 Version 2 (SF-36 v2) Score | Baseline, Week 64
Change from Baseline in EQ-5D-5L | Baseline, Week 64
Change from Baseline in Control of Eating Questionnaire (CoEQ) Score | Baseline, Week 64
Achievement of Improved Categorical Shift in Patient Global Improvement of Status (PGIS) Physical Function Weight | Baseline, Week 64
Change in Medication Use | Baseline through Week 64
Percent Change from Baseline in Body Weight in Participants with Prediabetes at Randomization | Baseline, Week 168
Pharmacokinetics (PK): Maximum Concentration at Steady State (Cmax,ss) | Baseline through Week 64
PK: Area Under the Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-ᴛ)ss) | Baseline through Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (172):
- United States (42):
  - MFA Clinical Research, Tuscaloosa, Alabama
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Neighborhood Healthcare Institute of Health, Escondido, California
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Care Access - Sacramento, Sacramento, California
  - Southern California Clinical Research, Santa Ana, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - BioMed Research & Medical Center, Miami, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - AHF Pensacola, Pensacola, Florida
  - IMA Clinical Research St. Petersburg, St. Petersburg, Florida
  - Teak Research Consults - Dunwoody, Dunwoody, Georgia
  - Teak Research Consults, Lawrenceville, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Care Access - Lake Charles (Bayou Pines), Lake Charles, Louisiana
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - MedStar Health Research Institute (MedStar Physician Based Research Network), Hyattsville, Maryland
  - Care Access - Quincy, Quincy, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - AMR Clinical, Las Vegas, Nevada
  - IMA Clinical Research Warren, Warren Township, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Rochester Clinical Research, LLC, Rochester, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Accellacare - Mt Pleasant, Mt. Pleasant, South Carolina
  - AMR Clinical, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Bellaire, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Discovery Clinical Trials - San Antonio, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - AMR Clinical, Norfolk, Virginia
- Argentina (17):
  - CONEXA Investigacion Clinica S.A., Buenos Aires
  - CIPREC, Buenos Aires
  - Cardiología Palermo, Buenos Aires
  - Glenny Corp. S.A., Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - CEDIC, CABA
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - CIPADI - Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz
  - INECO Neurociencias Oroño, Rosario
  - Instituto Especialidades de la Salud Rosario, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Laboratorio de Hemostasia y Trombosis, Rosario
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - Centro Modelo de Cardiología, San Miguel de Tucumán
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
- Australia (13):
  - Emeritus Research, Botany
  - Core Research Group, Brisbane
  - Paratus Clinical Research Canberra, Bruce
  - Emeritus Research, Camberwell
  - Life Clinical Research, Ipswich
  - Paratus Clinical Research Central Coast, Kanwal
  - University of the Sunshine Coast (UniSC) Clinical Trials - Meadowbrook, Meadowbrook
  - Momentum Sunshine, Melbourne
  - Paratus Clinical Research - Melbourne, Melbourne
  - AIM Research, Merewether
  - Fusion Clinical Research, Norwood
  - USC Clinical Trials Sunshine Coast, Sippy Downs
  - Brecken Health Bunbury, South Bunbury
- Belgium (4):
  - ANIMA Research, Alken
  - Jessa Ziekenhuis, Hasselt
  - Kormont, Kluisbergen
  - Gezondheidshuis De Gloed, Machelen
- Brazil (13):
  - Chronos Pesquisa Clínica, Brasília
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Sao Lucas, Campinas
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - IBPClin - Instituto Brasil de Pesquisa Clínica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali), São Paulo
  - CPCLIN, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - CEDOES, Vitória
  - Integral Pesquisa e Ensino, Votuporanga
- Canada (9):
  - Aggarwal and Associates Limited, Brampton
  - Med Trust Research, Courtice
  - Dawson Clinical Research Inc., Guelph
  - Winterberry Research Inc., Hamilton
  - The Wharton Medical Clinic Clinical Trials Inc, Hamilton
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
  - Bluewater Clinical Research Group Inc., Sarnia
  - Diex Recherche Inc. Division Trois-Rivieres, Trois-Rivières
- China (13):
  - Luhe Hospital, Beijing
  - Beijing Pinggu District Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Zhujiang Hospital, Guangzhou
  - The Second People's Hospital of Hefei, Hefei
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - Jiangsu Province Official Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - Shanghai Sixth People's Hospital, Shanghai
- Germany (13):
  - Zentrum fur klinische Forschung - Köln, Cologne
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - StudyPoint Duisburg, Duisburg
  - InnoDiab Forschung Gmbh, Essen
  - Medizentrum Essen Borbeck, Essen
  - Diabetes Zentrum Wilhelmsburg, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
  - AmBeNet GmbH, Leipzig
  - Diabetologische Schwerpunktpraxis Dr. Staudenmeyer & Dr. Schiwietz, Lingen
  - BAG Drs. Med. Quist PartG, Mainz
  - CRS Clinical Research Services Mannheim, Mannheim
  - RED-Institut GmbH, Oldenburg
  - Praxis Sauter & Sauter & Vorbach, Wangen
- India (10):
  - Endolife Speciality Hospitals, Guntur
  - Gauhati Medical College and Hospital, Guwahati
  - Care Hospitals Hyderabad- Banjara Hills, Hyderabad
  - Mandya Institute Of Medical Sciences, Mandya
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai
  - Mysore Medical College, Mysore
  - All India Institute of Medical Sciences (AIIMS) - Nagpur, Nagpur
  - Supe Heart & Diabetes Hospital and Research Centre, Nashik
  - Lifepoint Multispeciality Hospital, Pune
  - Prabhu Diabetes Multi-Speciality Centre, Trichy
- Japan (9):
  - Adachi Kyosai Hospital, Adachi-ku
  - Nihonbashi Sakura Clinic, Chūōku
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chūōku
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Boocs Clinic Fukuoka, Fukuoka
  - Patient First Clinic Ginza-Shimbashi, Minato
  - Kanno Naika, Mitaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi
  - Higashi Shinjuku Clinic, Tokyo
- Poland (9):
  - Zdrowie Osteo-Medic, Bialystok
  - Legeartis - Poradnie Specjalistyczne, Bialystok
  - Medyczne Centrum Diabetologiczno Endokrynologiczno Metaboliczne DIAB-ENDO-MET, Krakow
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Gabinety TERPA, Lublin
  - Ekamed, Lublin
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Pracownia Badań Klinicznych Salus, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 SUM, Zabrze
- Puerto Rico (2):
  - Puerto Rico Health and Wellness Institute, Dorado
  - Wellness clinical Research Vega Baja, Vega Baja
- South Korea (5):
  - Gachon University Gil Medical Center, Namdong-gu
  - Konyang University Hospital, Seogu
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Taiwan (5):
  - Chiayi Christian Hospital, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (8):
  - Layton Medical Centre, Blackpool
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Ashton Medical Group - Chapel House, Lancashire
  - Royal Lancaster Infirmary, Lancaster
  - Altnagelvin Area Hospital, Londonderry
  - Wansford Research Limited, Peterborough
  - Abbeywell Surgery, Romsey
  - Rame Group Practice, Torpoint

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/